CLINICAL TRIAL: NCT03130270
Title: Phase II Trial of Maintenance Apatinib After Second-Line Treatment for Locally Recurrent or Metastatic Nasopharyngeal Carcinoma
Brief Title: Maintenance Treatment of Apatinib in Nasopharyngeal Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Guilin Medical University, China (Other)
Collaborators: Wuzhou Red Cross Hospital (Other); Guangxi Naxishan Hospital (Other); People's Hospital of Guangxi Zhuang Autonomous Region (Other)
Responsible Party: Principal Investigator, Wei Jiang, Guilin Medical University, Guilin Medical University, China
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GLMU-02
Record Dates: First submitted 2017-04-21; First posted 2017-04-26 (Actual); Last update posted 2018-05-16 (Actual); Status verified 2018-05

CONDITIONS: Nasopharyngeal Carcinoma
Keywords: nasopharyngeal carcinoma; disease-free survival; adverse reaction
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — apatinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Apatinib group (Experimental): Apatinib mesylate tablet：the starting dose was 500 mg, orally, qd; tolerance assessment for a cycle, patients with poorly tolerance were treated with low dose (500 mg, qd), and patients with well tolerance were treated with high dose (750 mg, qd).
  Interventions: Drug: Apatinib mesylate tablet

INTERVENTIONS:
Drug: Apatinib mesylate tablet — Patients with locally recurrent or metastatic nasopharyngeal carcinoma (NPC) after second-line treatment are assigned to receive apatinib mesylate tablet. A treatment cycle was defined as 28 days (4 weeks). The starting dose was 500 mg, orally, qd; tolerance assessment for a cycle, patients with poorly tolerance were treated with low dose (500 mg, qd), and patients with well tolerance were treated with high dose (750 mg, qd). All patients continuous treatment until progression disease or non-tolerated toxicity.
  Note: good tolerance was defined that no grade 3/4 hematology or/and non hematologic side effects occurred within 4 weeks after initiation treatment; poor tolerance was defined that grade 3/4 hematology or/and non hematologic side effects appeared within 4 weeks after initiation treatment.
  Other Names: No.

SUMMARY:
The study is to evaluate the efficacy and safety of Apatinib for later treatment of patients(after second-line treatment for locally recurrent or metastatic nasopharyngeal carcinoma), including overall survival (OS), distant metastasis-free survival (DMFS) and locoregional relapse-free survival (LRRFS); the relationship between EBV DNA copy number and survival after radiotherapy or radiochemotherapy; Quality of life score (QoL); evaluation of drug safety.

DETAILED DESCRIPTION:
In locally advanced nasopharyngeal carcinoma(NPC), although fist-line therapy with radiotherapy and chemotherapy (Cisplatin/Docetaxel/5-Fu) and second-line therapy with chemotherapy has been given, patients still locally recurrence and distant metastasis. There is no standard treatment recommendation for locally recurrent or metastatic NPC who failed to second-line therapy. Apatinib has been approved as a second-line treatment for advanced gastric cancer. Several phase III studies of liver cancer, non small cell lung cancer and other tumors also showed apatinib has less toxicities and better tolerance. However, the clinical application of apatinib in nasopharyngeal carcinoma is still lack of evidence-based medicine. And this trial is designed to investigate the efficacy and safety of apatinib in locally recurrent or metastatic NPC.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients aged ranging from 18 to 70 years old.
2. Patients with newly histologically proven nasopharyngeal carcinoma (NPC).
3. Local recurrent NPC patients after comprehensive treatment, including clinical examination found a clear local area residue: electronic nasopharyngoscope found clear residual or enlarged cervical lymph nodes.
4. Distant metastatic NPC patients after comprehensive treatment, including liver B ultrasound, chest X-ray, bone scan or other clinicians consider appropriate tests such as CT, MRI or PET/CT found distant metastases.
5. Comprehensive treatment of local recurrence or distant metastasis after line or second-line therapy found progressive disease.
6. Eastern Cooperative Oncology Group (ECOG) performance status of 0 - 1.
7. Patient who has the expected survival time more than 3 months.
8. Adequate hematological function: hemoglobin >80 g/L (no transfusion within 14 days), neutrophil count > 1.5×109/L, platelet count 80×109/L.
9. Adequate liver function (serum total bilirubin ≤ 1.5 mg/dL, serum transminase ≤ 2.5 times higher than upper limit).
10. Adequate renal function (creatinine clearance ≥ 50 mL/min).
11. Participants volunteered to participate in this study, signed informed consent, good compliance and cooperated with us to complete the follow-up.

Exclusion Criteria:

1. Before treatment, MRI showed that the tumor might be an important risk factor (for example, wrapping around the internal carotid artery / vein); or researchers judged that the tumor is a high risk of serious blood vessel bleeding during the treatment.
2. Patient who has serious hemorrhages, any serious bleeding events classification at 3 degree or more (according to CTCAE4.0) within the last 4 weeks.
3. Patient who has high blood pressure can not be controlled by a single antihypertensive drug treatment (Systolic pressure > 140 mmHg, diastolic pressure > 90 mmHg); any unstable angina pectoris; with a history of angina pectoris were newly diagnosed with angina pectoris within 3 months before screening; any myocardial infarction events occurred within 6 months before screening; arrhythmia (including QTcF: male ≥ 450ms, female ≥ 470 ms) need long time use of antiarrhythmic drugs and heart function insufficiency ≥II according to New York Heart Association class.
4. Patient who has positive urine protein.
5. Patient who has abnormal coagulation and bleeding tendency (signed informed consent before 14 days, and must be satisfied: INR is in the normal range without the use of anticoagulants); Application of anticoagulants or vitamin K antagonists such as Hua Falin, heparin or its analogues, with international normalized ratio (INR) is less than 1.5, allows the use of small dose Hua Falin (1 mg orally, once daily) or small dose aspirin (total dose ≤ 100 mg daily).
6. Medical history of arteriovenous thrombosis event within the past year, such as cerebral vascular accident (including transient ischemic attack) and deep venous thrombosis (venous catheter thrombosis caused by chemotherapy and investigator judged that the patient had recovered, these patients should be except) and pulmonary embolism.
7. A healed wound for long time or incomplete fracture.
8. Any factors that affect the oral drug, such as the inability to swallow, diarrhea and intestinal obstruction.
9. For females: patients should be surgical sterilization or postmenopausal patients, or willing to receive a medical approved contraception during treatment and 6 months after the end of the treatment; serum or urine pregnancy test must be negative, and must be non lactating period within 7 days before study; for males: patients should be treated with surgical sterilization or willing to receive a medical approved contraception during treatment and 6 months after the end of the treatment.
10. History of psychotropic substance abuse and can not be removed or psychiatric disorders.
11. Medical history of immunodeficiency, or other acquired, congenital immunodeficiency disease, or history of organ transplantation.
12. Any serious harm to the subject's safety or evidence of significant medical illness that in the investigator's judgment will substantially increase the risk associated with the subject's participation in and completion of the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2019-04-08 (Estimated); Study Completion 2019-12-08 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) after Second-Line Treatment for Locally Recurrent or Metastatic Nasopharyngeal Carcinoma | up to 24 months
  To evaluate ORR every 6-8 weeks after initiation of apatinib.

SECONDARY OUTCOMES:
Disease-free survival (DFS) | up to 24 months
  The time from the first day of therapy to locoregional relapse, distant relapse again or tumor-related death.
Overall survival (OS) | up to 24 months
  The time from the first day of therapy to death or last follow-up.
Toxicity evaluation | up to 24 months
  Related toxicities were assessed using the National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) Version 4.0.

CONTACTS AND LOCATIONS:
Overall Officials: Wei Jiang, Principal Investigator — Guilin Medical University
Locations (4):
- China (4):
  - Guilin Medical University, Guilin, Guangxi
  - Nanxishan hospital, Guilin, Guangxi
  - National Hospital of Guangxi Zhuang Autonomous Region, Nanning, Guangxi
  - Wuzhou Red Cross Hospital, Wuzhou, Guangxi

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ruan X, Liang JH, Pan Y, Cai R, Zhang RJ, He Z, Yang X, Niu Z, Jiang W. Apatinib for the treatment of metastatic or locoregionally recurrent nasopharyngeal carcinoma after failure of chemotherapy: A multicenter, single-arm, prospective phase 2 study. Cancer. 2021 Sep 1;127(17):3163-3171. doi: 10.1002/cncr.33626. Epub 2021 May 27. PMID 34043812